CLINICAL TRIAL: NCT03903159
Title: Addiction Recovery in a Rural Minnesota Community: Piloting "Positive Peer Journaling" Part II
Brief Title: Piloting "Positive Peer Journaling" a Journaling Practice to Support Recovery From Addiction
Acronym: PPJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004619
Record Dates: First submitted 2019-01-18; First posted 2019-04-04 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Other): Positive Peer Journaling (PPJ)
  Interventions: Behavioral: Positive Peer Journaling (PPJ)

INTERVENTIONS:
Behavioral: Positive Peer Journaling (PPJ) — PPJ is a journaling practice to support addiction recovery. PPJ encourages past 24 hour review and upcoming 24 hour planning to improve quality of life in recovery and reduce relapse. PPJ uses standard lined journals with column headings under which individuals make bullet-pointed lists. On the left hand page, past 24 hours is recalled, itemizing "good" and "bad" things that happened and things for which one is grateful. Wishes for others are also expressed on this page. On the right hand page, values-based activities for the upcoming 24 hours are planned via headings representing valued life domains such as "recovery," "work/school," "spirituality," "home and household," and "health."

SUMMARY:
The main objective of this study is development of the Positive Peer Journaling (PPJ) intervention and the feasibility, acceptability, and logistics of treatment delivery. A second objective is to observe whether PPJ is associated with improvement in hypothesized outcomes. The primary outcomes the investigators will examine are enhanced treatment retention and reduced recurrence of substance use. The investigators will also explore the association between the intervention and a set of hypothesized mediators of the effect of the intervention on outcomes, e.g., improvement in mood and satisfaction with recovery.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years of age,
* meet DSM-V criteria for past-year SUD as primary or secondary diagnosis,
* English literacy sufficient to make short written lists needed to complete PPJ and homework assessments,
* minimum 2 weeks sustained abstinence,
* completed first 2 weeks of treatment at Wayside (approximately 2 weeks), a residential substance use disorder treatment program and the recruitment site,
* priority will go to participants who are from or moving back to a rural area or small town defined as a population less than 10,500,
* agree to be audio recorded in group meetings and in individual meetings with research staff,
* currently are clients in the Wayside residential program,
* participants must be English speaking and literacy must be strong enough to write short lists and to understand the questions asked in the questionnaires.
* Priority will go to women who will be residing at Wayside for the duration of the study activities (and not moving out after one week, for example).

Exclusion Criteria:

* presence of a psychotic disorder, psychiatric condition (e.g., suicidal ideation), or cognitive impairment (e.g., severe dementia, traumatic brain injury) limiting ability to give consent and/or participate in the study;
* severe psychiatric illness (current schizophrenia, major depression with suicidal ideation);
* personality disorders that would interfere with satisfactory participation in or completion of the study protocol,
* inability to give informed, voluntary consent to participate,
* lack of sufficient English literacy to participate, defined as inability to make a list of 5 things they did yesterday and inability to understand questionnaire items,
* any impairment, activity, or situation that in the judgement of the research staff would prevent satisfactory participation in or completion of the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The host setting is a residential substance use disorder treatment facility the serves only women.
Enrollment: 15 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Krentzman, Principal Investigator — University of Minnesota
Locations (1):
- Wayside Women's Treatment Center, Saint Louis Park, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 15
Completed | 10
Not Completed | 5
Not completed — Discharged with Staff Approval | 2
Not completed — Discharged at Staff Request | 2
Not completed — Discharged Against Staff Advice | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Treatment Retention
Description: Percentage of participants who were retained in treatment at the host facility until the end of the study or who left the residential treatment facility on good terms during the course of the study.
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
percentage of participants | 73.3

2. Primary Outcome: Substance Use
Description: Evidence that the individual used drugs or alcohol during the intervention period. This will be assessed via positive drug screen (urine test or breathalizer) or participant self-report of substance use. Reported as the number of participants who use illicit substances during the study.
Time Frame: 8 weeks
Measure: Number; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 4

3. Primary Outcome: Percentage of Group Sessions Attended
Description: Percentage of group sessions will be calculated by taking the number of group sessions attended divided by total number of group sessions offered. Outcome is reported as the overall percentage of group attendance for all 15 participants combined.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percent of sessions attended
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
percent of sessions attended | 78.3 (26.5)

4. Primary Outcome: Number of PPJ Journal Entries Made
Description: Total count of the number of PPJ journal entries made over the course of the study
Time Frame: 8 weeks
Measure: Number; unit: number of journal entries
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
number of journal entries | 196

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT03903159/Prot_SAP_000.pdf